CLINICAL TRIAL: NCT00829166
Title: A Randomized, Multicenter, Phase III Open-label Study of the Efficacy and Safety of Trastuzumab MCC-DM1 vs. Capecitabine + Lapatinib in Patients With HER2-Positive Locally Advanced or Metastatic Breast Cancer Who Have Received Prior Trastuzumab-Based Therapy
Brief Title: A Study of Trastuzumab Emtansine Versus Capecitabine + Lapatinib in Participants With HER2-positive Locally Advanced or Metastatic Breast Cancer
Acronym: EMILIA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BO21977; TDM4370g (Other: Genentech)
Record Dates: First submitted 2009-01-22; First posted 2009-01-26 (Estimated); Results first posted 2013-04-23 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Ado-Trastuzumab Emtansine; Lapatinib; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Trastuzumab emtansine (Experimental): Participants will receive trastuzumab emtansine 3.6 milligrams per kilogram (mg/kg) intravenous (IV) infusion over 30-90 minutes on Day 1 of each 21-day treatment cycle until disease progression (PD) (as assessed by the investigator), unmanageable toxicity, or study termination.
  Interventions: Drug: Trastuzumab emtansine
- Lapatinib + Capecitabine (Active Comparator): Participants will receive lapatinib 1250 mg (five 250 mg tablets) orally once daily during each 21-day cycle + capecitabine 1000 milligrams per square meter (mg/m^2) orally twice daily on Days 1-14 of each 21-day treatment cycle until PD (as assessed by the investigator), unmanageable toxicity, or study termination. Eligible participants will cross over to receive trastuzumab emtansine if second interim analysis demonstrates statistically significant overall survival benefit in favor of trastuzumab emtansine.
  Interventions: Drug: Lapatinib; Drug: Capecitabine

INTERVENTIONS:
Drug: Trastuzumab emtansine — Trastuzumab emtansine 3.6 mg/kg IV infusion over 30-90 minutes on Day 1 of each 21-day treatment cycle.
  Other Names: T-DM1; Trastuzumab-MCC-DM1; RO5304020
  Arms: Trastuzumab emtansine
Drug: Lapatinib — Lapatinib 1250 mg (five 250 mg tablets) orally once daily during each 21-day cycle.
  Other Names: Tykerb; Tyverb
  Arms: Lapatinib + Capecitabine
Drug: Capecitabine — Capecitabine 1000 mg/m^2 orally twice daily on Days 1-14 of each 21-day treatment cycle.
  Other Names: Xeloda
  Arms: Lapatinib + Capecitabine

SUMMARY:
This is a Phase III, randomized, multicenter, international, 2-arm, open-label clinical trial designed to compare the safety and efficacy of trastuzumab emtansine (T-DM1) with that of capecitabine + lapatinib in participants with human epidermal growth factor receptor 2 (HER2)-positive locally advanced or metastatic breast cancer. Participants will be treated until disease progression (PD), unmanageable toxicity, or study termination. Once disease progression is reported, all participants will be followed for survival every 3 months until death, loss to follow-up, withdrawal of consent, or study termination.

ELIGIBILITY:
Inclusion Criteria:

* HER2 status must be prospectively, centrally tested and be HER2-positive based on central laboratory assay results
* Histologically or cytologically confirmed invasive breast cancer
* Prior treatment for breast cancer in the adjuvant, unresectable, locally advanced, or metastatic setting must include both a taxane, alone or in combination with another agent, and trastuzumab, alone or in combination with another agent
* Documented progression (which occur during or after most recent treatment or within 6 months after completing of adjuvant therapy) of incurable, unresectable, locally advanced or metastatic breast cancer, defined by the investigator
* Measurable and/or nonmeasurable disease; participants with central nervous system-only disease are excluded
* Cardiac ejection fraction greater than or equal to (>/=) 50 percent (%) by either echocardiogram or multi-gated acquisition scan
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* For women of childbearing potential and men with partners of childbearing potential, agreement to use a highly effective, non-hormonal form of contraception; contraception use should continue for the duration of the study treatment and for at least 6 months after the last dose of study treatment

Exclusion Criteria:

* History of treatment with trastuzumab emtansine
* Prior treatment with lapatinib or capecitabine
* Peripheral neuropathy of Grade >/= 3 per National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE), Version 3.0
* History of other malignancy within the last 5 years, except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, Stage 1 uterine cancer, synchronous or previously diagnosed HER2-positive breast cancer, or cancers with a similar curative outcome as those mentioned above
* History of receiving any anti-cancer drug/biologic or investigational treatment within 21 days prior to randomization except hormone therapy, which could be given up to 7 days prior to randomization; recovery of treatment-related toxicity consistent with other eligibility criteria
* History of radiation therapy within 14 days of randomization
* Brain metastases that are untreated, symptomatic, or require therapy to control symptoms, as well as any history of radiation, surgery, or other therapy, including steroids, to control symptoms from brain metastases within 2 months (60 days) of randomization
* History of symptomatic congestive heart failure or serious cardiac arrhythmia requiring treatment
* History of myocardial infarction or unstable angina within 6 months of randomization
* Current dyspnea at rest due to complications of advanced malignancy or current requirement for continuous oxygen therapy
* Current severe, uncontrolled systemic disease (for example, clinically significant cardiovascular, pulmonary, or metabolic disease)
* Pregnancy or lactation
* Current known active infection with human immunodeficiency virus (HIV), hepatitis B virus, or hepatitis C virus
* Presence of conditions that could affect gastrointestinal absorption: Malabsorption syndrome, resection of the small bowel or stomach, and ulcerative colitis
* History of intolerance (such as Grade 3-4 infusion reaction) to trastuzumab
* Known hypersensitivity to 5-fluorouracil or known dihydropyrimidine dehydrogenase deficiency
* Current treatment with sorivudine or its chemically related analogs, such as brivudine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 991 (Actual)
Dates: Start 2009-02; Primary Completion 2012-07 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (281):
- United States (152):
  - Chandler, Arizona
  - Tucson, Arizona
  - Anaheim, California
  - Bakersfield, California
  - Baldwin Park, California
  - Bellflower, California
  - Duarte, California
  - Fontana, California
  - Hayward, California
  - Irvine, California
  - La Jolla, California
  - La Mesa, California
  - Loma Linda, California
  - Long Beach, California
  - Los Angeles, California
  - Montebello, California
  - Newport Beach, California
  - Oakland, California
  - Panorama City, California
  - Riverside, California
  - Roseville, California
  - Sacramento, California
  - San Diego, California
  - San Francisco, California
  - San Jose, California
  - Santa Clara, California
  - Santa Maria, California
  - Santa Monica, California
  - South San Francisco, California
  - Thousand Oaks, California
  - Vallejo, California
  - Walnut Creek, California
  - Woodland Hills, California
  - Fort Collins, Colorado
  - Norwalk, Connecticut
  - Norwich, Connecticut
  - Stamford, Connecticut
  - Washington D.C., District of Columbia
  - Boca Raton, Florida
  - Fernandina Beach, Florida
  - Fort Lauderdale, Florida
  - Fort Myers, Florida
  - Hollywood, Florida
  - Jacksonville, Florida
  - Kissimmee, Florida
  - Lakeland, Florida
  - Miami, Florida
  - Orange Park, Florida
  - Pembroke Pines, Florida
  - Athens, Georgia
  - Atlanta, Georgia
  - Carrolton, Georgia
  - Cartersville, Georgia
  - Decatur, Georgia
  - Douglasville, Georgia
  - Macon, Georgia
  - Marietta, Georgia
  - Boise, Idaho
  - Meridian, Idaho
  - Nampa, Idaho
  - Post Falls, Idaho
  - Twin Falls, Idaho
  - Chicago, Illinois
  - Decatur, Illinois
  - Effingham, Illinois
  - Joliet, Illinois
  - Morris, Illinois
  - Peoria, Illinois
  - Skokie, Illinois
  - Zion, Illinois
  - Bettendorf, Iowa
  - Wichita, Kansas
  - Paducah, Kentucky
  - Covington, Louisiana
  - Lafayette, Louisiana
  - Marrero, Louisiana
  - Metairie, Louisiana
  - New Orleans, Louisiana
  - Kittery, Maine
  - Wells, Maine
  - York Village, Maine
  - Baltimore, Maryland
  - Bethesda, Maryland
  - Rockville, Maryland
  - Boston, Massachusetts
  - Burlington, Massachusetts
  - Peabody, Massachusetts
  - Brownstown, Michigan
  - Dearborn, Michigan
  - Detroit, Michigan
  - Saint Joseph, Michigan
  - West Bloomfield, Michigan
  - Edina, Minnesota
  - Maplewood, Minnesota
  - Minneapolis, Minnesota
  - Saint Louis Park, Minnesota
  - Saint Paul, Minnesota
  - City of Saint Peters, Missouri
  - Joplin, Missouri
  - Kansas City, Missouri
  - St Louis, Missouri
  - Missoula, Montana
  - Omaha, Nebraska
  - Henderson, Nevada
  - Cherry Hill, New Jersey
  - Hackensack, New Jersey
  - Morristown, New Jersey
  - Parsippany, New Jersey
  - Voorhees Township, New Jersey
  - Santa Fe, New Mexico
  - Brockport, New York
  - Canandaigua, New York
  - Fresh Meadows, New York
  - Geneva, New York
  - Greece, New York
  - Lake Success, New York
  - Mount Kisco, New York
  - Rochester, New York
  - Stony Brook, New York
  - Charlotte, North Carolina
  - Durham, North Carolina
  - Hickory, North Carolina
  - Kinston, North Carolina
  - Washington, North Carolina
  - Cleveland, Ohio
  - Columbus, Ohio
  - Middletown, Ohio
  - Newark, Ohio
  - Sandusky, Ohio
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - East Providence, Rhode Island
  - Columbia, South Carolina
  - North Charleston, South Carolina
  - Memphis, Tennessee
  - Nashville, Tennessee
  - Austin, Texas
  - Bryan, Texas
  - Cypress, Texas
  - Dallas, Texas
  - El Paso, Texas
  - Houston, Texas
  - Shenandoah, Texas
  - Temple, Texas
  - Fairfax, Virginia
  - Gig Harbor, Washington
  - Lakewood, Washington
  - Puyallup, Washington
  - Tacoma, Washington
  - Milwaukee, Wisconsin
  - Wausau, Wisconsin
- Bosnia and Herzegovina (2):
  - Banja Luka
  - Sarajevo
- Brazil (11):
  - Belo Horizonte
  - Curitiba
  - Goiânia
  - Itajaí
  - Jaú
  - João Pessoa
  - Porto Alegre
  - Porto Alegre - Rs
  - Rio de Janeiro
  - Santo André
  - São Paulo
- Bulgaria (3):
  - Plovdiv
  - Sofia
  - Varna
- Canada (10):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Kelowna, British Columbia
  - Vancouver, British Columbia
  - Halifax, Nova Scotia
  - Greater Sudbury, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
  - Greenfield Park, Quebec
  - Montreal, Quebec
- Colombia (2):
  - Bogotá
  - Montería
- Denmark (3):
  - Copenhagen
  - Herlev
  - Odense
- Finland (3):
  - Helsinki
  - Tampere
  - Turku
- France (11):
  - Avignon
  - Bordeaux
  - Brest
  - Caen
  - Dijon
  - La Roche-sur-Yon
  - Montpellier
  - Paris
  - Saint-Brieuc
  - Saint-Herblain
  - Vandœuvre-lès-Nancy
- Germany (11):
  - Aschaffenburg
  - Berlin
  - Bonn
  - Dortmund
  - Freiburg im Breisgau
  - Fürstenwalde
  - Hamburg
  - Karlsruhe
  - Kiel
  - Offenbach
  - Stralsund
- Hong Kong, Hong Kong
- India (5):
  - Bangalore
  - Gūrgaon
  - Kolkata
  - New Delhi
  - Pune
- Italy (14):
  - Aviano
  - Bologna
  - Candiolo
  - Genova
  - Meldola
  - Milan
  - Napoli
  - Negrar
  - Pisa
  - Reggio Emilia
  - Roma
  - Rozzano
  - Sassari
  - Terni
- Mexico (3):
  - Acapulco
  - Oaxaca City
  - Toluca
- New Zealand (2):
  - Newtown
  - Palmerston North
- Philippines (2):
  - Diliman, Quezon City
  - Quezon City, Luzon
- Poland (7):
  - Bialystok
  - Gdansk
  - Krakow
  - Lublin
  - Opole
  - Poznan
  - Warsaw
- Portugal (3):
  - Coimbra
  - Lisbon
  - Porto
- Russia (3):
  - Kemerovo
  - Moscow
  - Saint Petersburg
- Singapore, Singapore
- Ljubljana, Slovenia
- South Korea (2):
  - Kyunggi-do
  - Seoul
- Spain (8):
  - Barcelona
  - Córdoba
  - Lleida
  - Madrid
  - Santander
  - Seville
  - Valencia
  - Zaragoza
- Sweden (3):
  - Eskilstuna
  - Gaelve
  - Gothenburg
- Switzerland (2):
  - Lucerne
  - Sankt Gallen
- Taiwan (4):
  - Kaohsung
  - Taichung
  - Taipei
  - Taoyuan District
- United Kingdom (12):
  - Bournemouth
  - Cardiff
  - Denbigh
  - London
  - Manchester
  - New Castle Upon Tyne
  - Northwood
  - Poole
  - Preston
  - Romford
  - Sutton
  - Weston-super-Mare

REFERENCES:
- [Derived] Dieras V, Miles D, Verma S, Pegram M, Welslau M, Baselga J, Krop IE, Blackwell K, Hoersch S, Xu J, Green M, Gianni L. Trastuzumab emtansine versus capecitabine plus lapatinib in patients with previously treated HER2-positive advanced breast cancer (EMILIA): a descriptive analysis of final overall survival results from a randomised, open-label, phase 3 trial. Lancet Oncol. 2017 Jun;18(6):732-742. doi: 10.1016/S1470-2045(17)30312-1. Epub 2017 May 16. PMID 28526536
- [Derived] Verma S, Miles D, Gianni L, Krop IE, Welslau M, Baselga J, Pegram M, Oh DY, Dieras V, Guardino E, Fang L, Lu MW, Olsen S, Blackwell K; EMILIA Study Group. Trastuzumab emtansine for HER2-positive advanced breast cancer. N Engl J Med. 2012 Nov 8;367(19):1783-91. doi: 10.1056/NEJMoa1209124. Epub 2012 Oct 1. PMID 23020162
- [Derived] Scott AM, Wolchok JD, Old LJ. Antibody therapy of cancer. Nat Rev Cancer. 2012 Mar 22;12(4):278-87. doi: 10.1038/nrc3236. PMID 22437872

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants of "Lapatinib + Capecitabine" arm were allowed to cross over to receive trastuzumab emtansine based on statistically significant Overall Survival (OS) benefit in favor of trastuzumab emtansine demonstrated in second interim analysis (cut-off date 31 July 2012). The safety analysis of the arm was then reported.
Groups:
- Trastuzumab Emtansine: Participants received trastuzumab emtansine 3.6 milligrams per kilogram (mg/kg) intravenous (IV) infusion over 30-90 minutes on Day 1 of each 21-day treatment cycle until disease progression (PD) (as assessed by the investigator), unmanageable toxicity, or study termination.
- Lapatinib + Capecitabine: Participants received lapatinib 1250 mg (five 250 mg tablets) orally once daily during each 21-day cycle + capecitabine 1000 milligrams per square meter (mg/m^2) orally twice daily on Days 1-14 of each 21-day treatment cycle until PD (as assessed by the investigator), unmanageable toxicity, or study termination. Participants of this group were allowed to cross over to receive trastuzumab emtansine based on statistically significant OS benefit in favor of trastuzumab emtansine demonstrated in second interim analysis.
Period: Overall Study
Arm/Group | Trastuzumab Emtansine | Lapatinib + Capecitabine
Started | 495 | 496
Treated | 490 | 488
Completed | 0 | 0
Not Completed | 495 | 496
Not completed — Death | 305 | 333
Not completed — Lost to Follow-up | 5 | 4
Not completed — Physician's Decision | 4 | 3
Not completed — Subject's Decision | 41 | 55
Not completed — Sponsor's Decision | 137 | 98
Not completed — Reason Not Specified | 3 | 3

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all randomized participants on the basis of the treatment assigned at randomization.
Groups:
- Trastuzumab Emtansine: Participants received trastuzumab emtansine 3.6 mg/kg IV infusion over 30-90 minutes on Day 1 of each 21-day treatment cycle until PD (as assessed by the investigator), unmanageable toxicity, or study termination.
- Lapatinib + Capecitabine: Participants received lapatinib 1250 mg (five 250 mg tablets) orally once daily during each 21-day cycle + capecitabine 1000 mg/m^2 orally twice daily on Days 1-14 of each 21-day treatment cycle until PD (as assessed by the investigator), unmanageable toxicity, or study termination. Participants of this group were allowed to cross over to receive trastuzumab emtansine based on statistically significant OS benefit in favor of trastuzumab emtansine demonstrated in second interim analysis.
- Total: Total of all reporting groups
Arm/Group | Trastuzumab Emtansine | Lapatinib + Capecitabine | Total
Number analyzed (Participants) | 495 | 496 | 991
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.2 (11.0) | 53.2 (10.8) | 52.7 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 494 | 492 | 986
  Male | 1 | 4 | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With PD or Death as Assessed by an Independent Review Committee (IRC)
Description: PD was assessed by an IRC using modified Response Evaluation Criteria in Solid Tumors (RECIST). All measurable lesions up to a maximum of 5 per organ and 10 in total were identified as target lesions (TLs) and recorded at baseline. TLs should be selected on the basis of their size (those with the longest diameter) and their suitability for accurate repeated measurements either by imaging or clinically. A sum of the longest diameter for all TLs was calculated as baseline sum longest diameter (SLD). All other lesions (or sites of disease) should be identified as non-TLs and recorded at baseline. PD for TLs was defined as greater than or equal to (>/=) 20 percent (%) increase in SLD, taking as reference smallest SLD recorded since treatment started or appearance of 1 or more new lesions. PD for non-TLs was defined as appearance of 1 or more new lesions and/or unequivocal progression of existing non-TLs. Percentage of Participants with PD by IRC or death from any cause was reported.
Time Frame: From the date of randomization through the data cut-off date of 14 Jan 2012 (up to 2 years, 11 months)
Population: ITT population included all randomized participants on the basis of the treatment assigned at randomization.
Measure: Number; unit: percentage of participants
Arm/Group | Trastuzumab Emtansine | Lapatinib + Capecitabine
Number analyzed (Participants) | 495 | 496
percentage of participants | 53.5 | 61.3

2. Primary Outcome: Progression-free Survival (PFS) as Assessed by an IRC (Co-primary Endpoint)
Description: Tumor response was assessed by an IRC according to modified RECIST. All measurable lesions up to a maximum of 5 per organ and 10 in total were identified as TLs (on the basis of their size and their suitability for accurate repeated measurements either by imaging or clinically) and recorded at baseline. A sum of the longest diameter for all TLs was calculated as baseline SLD. All other lesions were identified as non-TLs and recorded at baseline. PD for TLs: >/= 20% increase in the SLD, taking as reference the smallest SLD recorded since treatment started or appearance of 1 or more new lesions. PD for non-TLs: appearance of 1 or more new lesions and/or unequivocal progression of existing non-TLs. PFS: time from randomization to first documented PD by IRC or death from any cause (whichever occurred earlier). The median duration of PFS was estimated using Kaplan-Meier method. The 95% confidence interval (CI) was computed using the method of Brookmeyer and Crowley.
Time Frame: From the date of randomization through the data cut-off date of 14 Jan 2012 (up to 2 years, 11 months)
Population: ITT population included all randomized participants on the basis of the treatment assigned at randomization.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Trastuzumab Emtansine | Lapatinib + Capecitabine
Number analyzed (Participants) | 495 | 496
Months | 9.6 [8.25 to 10.64] | 6.4 [5.68 to 7.06]
Statistical Analysis 1: Comparison: Trastuzumab Emtansine vs Lapatinib + Capecitabine; Analysis stratified by region of enrollment, number of prior chemotherapeutic regimens (0-1 or greater than [>] 1), and visceral/ non-visceral disease; Test type: Superiority or Other; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.650, 95% CI 2-sided [0.549 to 0.771] — HR (relative to Lapatinib + Capecitabine) was estimated by Cox regression

3. Primary Outcome: Percentage of Participants Who Died: Second Interim Analysis
Description: The percentage of participants who died from any cause was reported. The results are reported from second interim analysis, which deemed to be the confirmatory.
Time Frame: From the date of randomization through the data cut-off date of 31 Jul 2012 (up to 3 years, 5 months)
Population: ITT population included all randomized participants on the basis of the treatment assigned at randomization.
Measure: Number; unit: percentage of participants
Arm/Group | Trastuzumab Emtansine | Lapatinib + Capecitabine
Number analyzed (Participants) | 495 | 496
percentage of participants | 30.1 | 36.7

4. Primary Outcome: Overall Survival: Second Interim Analysis (Co-primary Endpoint)
Description: OS was defined as the time from the date of randomization to the date of death from any cause. The median duration of OS was estimated using Kaplan-Meier method. The 95% CI was computed using the method of Brookmeyer and Crowley. The results are reported from second interim analysis, which deemed to be the confirmatory.
Time Frame: From the date of randomization through the data cut-off date of 31 Jul 2012 (up to 3 years, 5 months)
Population: ITT population included all randomized participants on the basis of the treatment assigned at randomization.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Trastuzumab Emtansine | Lapatinib + Capecitabine
Number analyzed (Participants) | 495 | 496
Months | 30.9 [26.81 to 34.27] | 25.1 [22.74 to 27.96]
Statistical Analysis 1: Comparison: Trastuzumab Emtansine vs Lapatinib + Capecitabine; Analysis stratified by region of enrollment, number of prior chemotherapeutic regimens (0-1 or >1), and visceral/ non-visceral disease; Test type: Superiority or Other; p = 0.0006, Log Rank; Hazard Ratio (HR) = 0.682, 95% CI 2-sided [0.548 to 0.849] — HR (relative to Lapatinib + Capecitabine) was estimated by Cox regression

5. Primary Outcome: Percentage of Participants Who Died: Final Analysis
Description: The percentage of participants who died from any cause was reported. The results reported are from the final analysis. The final analysis is descriptive.
Time Frame: From the date of randomization through the data cut-off date of 31 Dec 2014 (up to 5 years, 11 months)
Population: ITT population included all randomized participants on the basis of the treatment assigned at randomization.
Measure: Number; unit: percentage of participants
Arm/Group | Trastuzumab Emtansine | Lapatinib + Capecitabine
Number analyzed (Participants) | 495 | 496
percentage of participants | 61.2 | 67.1

6. Primary Outcome: Overall Survival: Final Analysis
Description: OS was defined as the time from the date of randomization to the date of death from any cause. The median duration of OS was estimated using Kaplan-Meier method. The 95% CI was computed using the method of Brookmeyer and Crowley. The results reported are from the final analysis. The final analysis is descriptive.
Time Frame: From the date of randomization through the data cut-off date of 31 Dec 2014 (up to 5 years, 11 months)
Population: ITT population included all randomized participants on the basis of the treatment assigned at randomization.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Trastuzumab Emtansine | Lapatinib + Capecitabine
Number analyzed (Participants) | 495 | 496
Months | 29.9 [26.32 to 34.10] | 25.9 [22.74 to 28.32]
Statistical Analysis 1: Comparison: Trastuzumab Emtansine vs Lapatinib + Capecitabine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0003, Log Rank; Hazard Ratio (HR) = 0.749, 95% CI 2-sided [0.639 to 0.877] — HR (relative to Lapatinib + Capecitabine) was estimated by Cox regression

7. Primary Outcome: Percentage of Participants Who Were Alive at Year 1
Description: 1 year survival was defined as the percentage of participants alive 1 year after starting treatment. The results reported are from the final analysis.
Time Frame: Year 1
Population: ITT population included all randomized participants on the basis of the treatment assigned at randomization.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Trastuzumab Emtansine | Lapatinib + Capecitabine
Number analyzed (Participants) | 495 | 496
percentage of participants | 85.3 [82.15 to 88.54] | 78.9 [75.19 to 82.65]

8. Primary Outcome: Percentage of Participants Who Were Alive at Year 2
Description: 2 year survival was defined as the percentage of participants alive 2 years after starting treatment. The results reported are from the final analysis.
Time Frame: Year 2
Population: ITT population included all randomized participants on the basis of the treatment assigned at randomization.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Trastuzumab Emtansine | Lapatinib + Capecitabine
Number analyzed (Participants) | 495 | 496
percentage of participants | 59.6 [55.10 to 64.06] | 52.4 [47.81 to 57.08]

9. Secondary Outcome: Percentage of Participants With PD or Death as Assessed by the Investigator
Description: PD was assessed by the investigator using modified RECIST. All measurable lesions up to a maximum of 5 per organ and 10 in total were identified as TLs and recorded at baseline. A sum of the longest diameter for all TLs was calculated as baseline SLD. PD for TLs was defined as >/=20% increase in the SLD, taking as reference the smallest SLD recorded since treatment started or the appearance of 1 or more new lesions. PD for non-TLs was defined as appearance of 1 or more new lesions and/or unequivocal progression of existing non-TLs. The percentage of participants who died or experienced PD by Investigator was reported.
Time Frame: From the date of randomization through the data cut-off date of 14 Jan 2012 (up to 2 years, 11 months)
Population: ITT population included all randomized participants on the basis of the treatment assigned at randomization.
Measure: Number; unit: percentage of participants
Arm/Group | Trastuzumab Emtansine | Lapatinib + Capecitabine
Number analyzed (Participants) | 495 | 496
percentage of participants | 58.0 | 67.5

10. Secondary Outcome: PFS as Assessed by the Investigator
Description: Tumor response was assessed by the investigator according to modified RECIST. All measurable lesions up to a maximum of 5 per organ and 10 in total were identified as TLs and recorded at baseline. A sum of the longest diameter for all TLs was calculated as baseline SLD. PD for TLs was defined as >/=20% increase in the SLD, taking as reference the smallest SLD recorded since treatment started or the appearance of 1 or more new lesions. PD for non-TLs was defined as appearance of 1 or more new lesions and/or unequivocal progression of existing non-TLs. PFS was defined as the time from randomization to first documented PD by Investigator or death from any cause (whichever occurred earlier). The median duration of PFS was estimated using Kaplan-Meier method. The 95% CI was computed using the method of Brookmeyer and Crowley.
Time Frame: From the date of randomization through the data cut-off date of 14 Jan 2012 (up to 2 years, 11 months)
Population: ITT population included all randomized participants on the basis of the treatment assigned at randomization.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Trastuzumab Emtansine | Lapatinib + Capecitabine
Number analyzed (Participants) | 495 | 496
Months | 9.4 [7.49 to 10.78] | 5.8 [5.59 to 6.93]
Statistical Analysis 1: Comparison: Trastuzumab Emtansine vs Lapatinib + Capecitabine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.658, 95% CI 2-sided [0.560 to 0.774] — HR (relative to Lapatinib + Capecitabine) was estimated by Cox regression

11. Secondary Outcome: Percentage of Participants With Objective Response (OR) as Assessed by an IRC
Description: Tumor response was assessed by an IRC according to modified RECIST. OR was defined as the percentage of participants with a complete response (CR) or partial response (PR). All measurable lesions up to a maximum of 5 per organ and 10 in total were identified as TLs and recorded at baseline. A sum of the longest diameter for all TLs was calculated as baseline SLD. For TLs, a CR was defined as the disappearance of all TLs and a PR was defined as >/= 30% decrease in the SLD of TLs, taking as reference the baseline SLD. For non-TLs, a CR was defined as the disappearance of all non-TLs and a PR was defined as the persistence of 1 or more non-TLs. Confirmation of response at a consecutive tumor assessment at least 4 weeks apart was required. Participants without a post-baseline tumor assessment were considered non-responders. The percentage of participants with CR or PR by IRC was reported. The 95% CI was computed using Blyth-Still Casella exact CI method.
Time Frame: From the date of randomization through the data cut-off date of 14 Jan 2012 (up to 2 years, 11 months)
Population: ITT population included all randomized participants on the basis of the treatment assigned at randomization. Only participants with measurable disease at baseline were included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Trastuzumab Emtansine | Lapatinib + Capecitabine
Number analyzed (Participants) | 397 | 389
percentage of participants | 43.6 [38.6 to 48.6] | 30.8 [26.3 to 35.7]
Statistical Analysis 1: Comparison: Trastuzumab Emtansine vs Lapatinib + Capecitabine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0002, Mantel-Haenszel chi-squared test; Difference in Objective Response Rates = 12.7, 95% CI 2-sided [6.0 to 19.4] — The 95% CI for the difference in objective response rate (Trastuzumab emtansine minus Lapatinib + Capecitabine) was computed by using the approximate normal method

12. Secondary Outcome: Duration of Objective Response (DOR) as Assessed by an IRC
Description: Tumor response was assessed by an IRC according to modified RECIST. DOR was defined as the time from first documented OR to first documented PD or death from any cause, whichever occurred earlier. OR was defined as a CR or PR determined on 2 consecutive tumor assessments at least 4 weeks apart. For TLs, CR was defined as the disappearance of all TLs; PR was defined as >/=30% decrease in the SLD of TLs, taking as reference the baseline SLD; and PD was defined as >/=20% increase in the SLD, taking as reference the smallest SLD recorded since treatment started or the appearance of 1 or more new lesions. For non-TLs, CR was defined as the disappearance of all non-TLs; PR was defined as the persistence of 1 or more non-TLs; and PD was defined as appearance of 1 or more new lesions and/or unequivocal progression of existing non-TLs. The 95% CI was computed using the method of Brookmeyer and Crowley.
Time Frame: From the date of randomization through the data cut-off date of 14 Jan 2012 (up to 2 years, 11 months)
Population: ITT population included all randomized participants on the basis of the treatment assigned at randomization. Only participants with an objective response were included in the analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Trastuzumab Emtansine | Lapatinib + Capecitabine
Number analyzed (Participants) | 173 | 120
Months | 12.6 [8.38 to 20.76] | 6.5 [5.45 to 7.16]

13. Secondary Outcome: Percentage of Participants With Clinical Benefit as Assessed by an IRC
Description: Tumor response was assessed by an IRC according to modified RECIST. Participants were considered as experienced clinical benefit if they had an OR or maintained stable disease (SD) for at least 6 months from randomization. OR: CR or PR determined on 2 consecutive tumor assessments >/=4 weeks apart. For TLs, CR: disappearance of all TLs; PR: >/=30% decrease in the SLD of TLs, taking as reference the baseline SLD; PD: >/=20% increase in the SLD, taking as reference the smallest SLD recorded since treatment started or appearance of 1 or more new lesions; and SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD. For non-TLs, CR: disappearance of all non-TLs; PR/SD: persistence of 1 or more non-TLs; and PD: appearance of 1 or more new lesions and/or unequivocal progression of existing non-TLs. Participants without a post-baseline tumor assessment were considered non-responders. The 95% CI was computed using Blyth-Still Casella exact CI method.
Time Frame: From the date of randomization through the data cut-off date of 14 Jan 2012 (up to 2 years, 11 months)
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Trastuzumab Emtansine | Lapatinib + Capecitabine
Number analyzed (Participants) | 397 | 389
percentage of participants | 58.2 [53.3 to 63.1] | 44.2 [39.2 to 49.2]
Statistical Analysis 1: Comparison: Trastuzumab Emtansine vs Lapatinib + Capecitabine; Test type: Superiority or Other; Difference in Clinical Benefit Rate = 14, 95% CI 2-sided [7.0 to 20.9] — The 95% CI for the difference in clinical benefit rate (Trastuzumab emtansine minus Lapatinib + Capecitabine) was computed by using the normal approximation method

14. Secondary Outcome: Percentage of Participants With Treatment Failure
Description: Treatment failure was defined as discontinuation of treatment for any reason, including PD (per investigator review), treatment toxicity, or death from any cause. For "Lapatinib + Capecitabine" arm, a participant was considered as treatment failure only if both drugs were discontinued. For TLs, PD was defined as >/=20% increase in the SLD, taking as reference the smallest SLD recorded since treatment started or the appearance of 1 or more new lesions. For non-TLs, PD was defined as appearance of 1 or more new lesions and/or unequivocal progression of existing non-TLs. Percentage of participants with treatment failure was reported.
Time Frame: From the date of randomization through the data cut-off date of 14 Jan 2012 (up to 2 years, 11 months)
Population: ITT population included all randomized participants on the basis of the treatment assigned at randomization.
Measure: Number; unit: percentage of participants
Arm/Group | Trastuzumab Emtansine | Lapatinib + Capecitabine
Number analyzed (Participants) | 495 | 496
percentage of participants | 63.2 | 74.8

15. Secondary Outcome: Time to Treatment Failure
Description: Time to treatment failure was defined as the time from randomization to discontinuation of treatment for any reason, including PD (per investigator review), treatment toxicity, or death from any cause. For "Lapatinib + Capecitabine" arm, a participant was considered as treatment failure only if both drugs were discontinued with treatment failure date as the later of the 2 discontinuation dates. For TLs, PD was defined as >/=20% increase in the SLD, taking as reference the smallest SLD recorded since treatment started or the appearance of 1 or more new lesions. For non-TLs, PD was defined as appearance of 1 or more new lesions and/or unequivocal progression of existing non-TLs. The median time to treatment failure was estimated using Kaplan-Meier method. The 95% CI was computed using the method of Brookmeyer and Crowley.
Time Frame: From the date of randomization through the data cut-off date of 14 Jan 2012 (up to 2 years, 11 months)
Population: ITT population included all randomized participants on the basis of the treatment assigned at randomization.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Trastuzumab Emtansine | Lapatinib + Capecitabine
Number analyzed (Participants) | 495 | 496
Months | 7.9 [6.41 to 9.00] | 5.8 [5.52 to 6.31]
Statistical Analysis 1: Comparison: Trastuzumab Emtansine vs Lapatinib + Capecitabine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.703, 95% CI 2-sided [0.602 to 0.820] — HR (relative to Lapatinib + Capecitabine) was estimated by Cox regression

16. Secondary Outcome: Percentage of Participants With Symptom Progression
Description: Symptom progression was defined as the documentation of a >/= 5-point decrease from baseline in the scoring of responses as measured by the Functional Assessment of Cancer Therapy-for participants with Breast Cancer (FACT-B) questionnaire with the Trial Outcomes Index-Physical/Functional/Breast (TOI-PFB) subscale. The FACT-B TOI-PFB subscale contained 24 items from 3 subsections of the FACT-B questionnaire: Physical well-being, functional well-being, and additional concerns for breast cancer participants (breast cancer subscale [BCS]). All items in the questionnaire were rated by the participant on a 5-point scale ranging from 0 ("not at all") to 4 ("very much"). The total score ranged from 0 to 96 with higher score indicating better perceived quality of life. The percentage of participants with symptom progression was reported.
Time Frame: From the date of randomization through the data cut-off date of 14 Jan 2012 (up to 2 years, 11 months)
Population: ITT population included all randomized participants on the basis of the treatment assigned at randomization. Only female participants with a Baseline assessment and at least 1 follow-up assessment were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Trastuzumab Emtansine | Lapatinib + Capecitabine
Number analyzed (Participants) | 450 | 445
percentage of participants | 54.7 | 57.8

17. Secondary Outcome: Time to Symptom Progression
Description: Time to symptom progression was defined as the time from randomization to the first documentation of a >/= 5-point decrease from baseline in the scoring of responses as measured by the FACT-B questionnaire with the TOI-PFB subscale. The FACT-B TOI-PFB subscale contained 24 items from 3 subsections of the FACT-B questionnaire: Physical well-being, functional well-being, and additional concerns for breast cancer participants (BCS). All items in the questionnaire were rated by the participant on a 5-point scale ranging from 0 ("not at all") to 4 ("very much"). The total score ranged from 0 to 96 with higher score indicating better perceived quality of life. The median time to symptom progression was estimated using Kaplan-Meier method. The 95% CI was computed using the method of Brookmeyer and Crowley.
Time Frame: From the date of randomization through the data cut-off date of 14 Jan 2012 (up to 2 years, 11 months)
Population: as for outcome 16
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Trastuzumab Emtansine | Lapatinib + Capecitabine
Number analyzed (Participants) | 450 | 445
Months | 7.1 [5.59 to 8.44] | 4.6 [4.14 to 5.78]
Statistical Analysis 1: Comparison: Trastuzumab Emtansine vs Lapatinib + Capecitabine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0121, Log Rank; Hazard Ratio (HR) = 0.796, 95% CI 2-sided [0.667 to 0.951] — HR (relative to Lapatinib + Capecitabine) was estimated by Cox regression

ADVERSE EVENTS:
Time Frame: Only study-related serious adverse events (SAEs) were reported from randomization to first treatment; all SAEs and non-SAEs were reported from start of treatment until 30 days after treatment; and thereafter only treatment related SAEs were reported until data cut-off date of 21-Sep-2015 (up to 6 years and 7 months). For participants who crossed over from lapatinib + capecitabine to trastuzumab emtansine, data is reported from time of cross-over until 21-Sep-2015 (up to 3 years and 2 months).
Description: Safety population included participants who received at least 1 dose of study medication. Safety analyses were based on the actual treatment received.
Groups:
- Lapatinib + Capecitabine/ Trastuzumab Emtansine: Participants of "Lapatinib + Capecitabine" arm were allowed to cross over to receive trastuzumab emtansine based on statistically significant OS benefit in favor of trastuzumab emtansine demonstrated in second interim analysis.
Arm/Group | Trastuzumab Emtansine | Lapatinib + Capecitabine | Lapatinib + Capecitabine/ Trastuzumab Emtansine
Serious Adverse Events (participants affected / at risk) | 92/490 | 99/488 | 19/136
Other Adverse Events (participants affected / at risk) | 474/490 | 471/488 | 115/136
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab Emtansine (N=490) | Lapatinib + Capecitabine (N=488) | Lapatinib + Capecitabine/ Trastuzumab Emtansine (N=136)
Unmapped (Bacteremia due to infected port) (Infections and infestations) | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0
Anaemia of malignant disease (Blood and lymphatic system disorders) | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 1 | 1
Angina pectoris (Cardiac disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 2 | 0
Pericarditis (Cardiac disorders) | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0
Macular hole (Eye disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 4 | 3 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 17 | 0
Enteritis (Gastrointestinal disorders) | 0 | 1 | 0
Fistula of small intestine (Gastrointestinal disorders) | 0 | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0 | 0
Gastrointestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 2 | 0
Intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 3 | 0
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 7 | 10 | 0
Malaise (General disorders) | 1 | 0 | 0
Asthenia (General disorders) | 1 | 2 | 1
Chest pain (General disorders) | 2 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 1 | 0
Multi-organ failure (General disorders) | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0
Pain (General disorders) | 2 | 1 | 0
Pyrexia (General disorders) | 8 | 3 | 2
Cholangitis (Hepatobiliary disorders) | 1 | 0 | 0
Cholangitis acute (Hepatobiliary disorders) | 0 | 0 | 1
Cholestasis (Hepatobiliary disorders) | 0 | 1 | 0
Hepatitis toxic (Hepatobiliary disorders) | 1 | 0 | 0
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 2 | 0
Nodular regenerative hyperplasia (Hepatobiliary disorders) | 0 | 0 | 1
Portal hypertension (Hepatobiliary disorders) | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 1 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0
Catheter site infection (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 2 | 3 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 1 | 0
Device related infection (Infections and infestations) | 2 | 0 | 0
Enterococcal infection (Infections and infestations) | 1 | 0 | 1
Erysipelas (Infections and infestations) | 0 | 1 | 0
Gastroenteritis norovirus (Infections and infestations) | 1 | 0 | 0
H1N1 influenza (Infections and infestations) | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0
Infection (Infections and infestations) | 0 | 1 | 0
Listeriosis (Infections and infestations) | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0
Neutropenic sepsis (Infections and infestations) | 2 | 0 | 0
Parotitis (Infections and infestations) | 1 | 0 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 4 | 1 | 1
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 0
Post procedural infection (Infections and infestations) | 0 | 1 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 2
Salmonellosis (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 1 | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0 | 0
Tooth infection (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 3 | 0 | 1
Urosepsis (Infections and infestations) | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Delayed haemolytic transfusion reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0
Extradural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 3 | 2 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0 | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0
Synovial rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wound (Injury, poisoning and procedural complications) | 1 | 0 | 0
Wound secretion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 2 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Spondylitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lentigo maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Second primary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 1 | 0
Coma (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 2 | 2 | 0
Epilepsy (Nervous system disorders) | 1 | 1 | 0
Headache (Nervous system disorders) | 1 | 2 | 0
Hemiplegia (Nervous system disorders) | 1 | 0 | 0
Hydrocephalus (Nervous system disorders) | 0 | 1 | 0
Metabolic encephalopathy (Nervous system disorders) | 1 | 0 | 0
Parkinson's disease (Nervous system disorders) | 1 | 0 | 0
Status epilepticus (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 2 | 0
Agitation (Psychiatric disorders) | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 1 | 0
Depression (Psychiatric disorders) | 0 | 2 | 0
Substance-induced psychotic disorder (Psychiatric disorders) | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 0
Ureteric obstruction (Renal and urinary disorders) | 0 | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1 | 0
Menometrorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 2 | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Alveolitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 9 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Abortion induced (Surgical and medical procedures) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 2 | 0
Labile blood pressure (Vascular disorders) | 1 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 2 | 0
Venous thrombosis (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab Emtansine (N=490) | Lapatinib + Capecitabine (N=488) | Lapatinib + Capecitabine/ Trastuzumab Emtansine (N=136)
Anaemia (Blood and lymphatic system disorders) | 67 | 40 | 11
Neutropenia (Blood and lymphatic system disorders) | 37 | 43 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 150 | 13 | 23
Dry eye (Eye disorders) | 0 | 0 | 7
Abdominal pain (Gastrointestinal disorders) | 43 | 50 | 0
Abdominal pain upper (Gastrointestinal disorders) | 60 | 45 | 0
Constipation (Gastrointestinal disorders) | 139 | 59 | 22
Diarrhoea (Gastrointestinal disorders) | 123 | 385 | 20
Dry mouth (Gastrointestinal disorders) | 85 | 26 | 20
Dyspepsia (Gastrointestinal disorders) | 51 | 57 | 7
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 8
Nausea (Gastrointestinal disorders) | 202 | 224 | 35
Stomatitis (Gastrointestinal disorders) | 20 | 70 | 0
Vomiting (Gastrointestinal disorders) | 98 | 145 | 13
Influenza like illness (General disorders) | 26 | 9 | 13
Asthenia (General disorders) | 91 | 86 | 23
Chest pain (General disorders) | 40 | 27 | 0
Chills (General disorders) | 42 | 16 | 13
Fatigue (General disorders) | 180 | 145 | 30
Mucosal inflammation (General disorders) | 33 | 93 | 0
Oedema peripheral (General disorders) | 38 | 38 | 10
Pain (General disorders) | 35 | 14 | 0
Pyrexia (General disorders) | 95 | 43 | 18
Hyperbilirubinaemia (Hepatobiliary disorders) | 13 | 46 | 0
Nasopharyngitis (Infections and infestations) | 50 | 41 | 14
Paronychia (Infections and infestations) | 2 | 59 | 0
Upper respiratory tract infection (Infections and infestations) | 56 | 40 | 14
Urinary tract infection (Infections and infestations) | 52 | 21 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 8
Alanine aminotransferase increased (Investigations) | 92 | 48 | 14
Aspartate aminotransferase increased (Investigations) | 123 | 53 | 25
Blood alkaline phosphatase increased (Investigations) | 26 | 23 | 9
Blood bilirubin increased (Investigations) | 21 | 32 | 11
Platelet count decreased (Investigations) | 0 | 0 | 8
Weight decreased (Investigations) | 38 | 37 | 7
Decreased appetite (Metabolism and nutrition disorders) | 105 | 117 | 21
Dehydration (Metabolism and nutrition disorders) | 9 | 25 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 47 | 45 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 102 | 46 | 21
Back pain (Musculoskeletal and connective tissue disorders) | 78 | 63 | 9
Bone pain (Musculoskeletal and connective tissue disorders) | 34 | 20 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 39 | 22 | 8
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 46 | 22 | 10
Myalgia (Musculoskeletal and connective tissue disorders) | 70 | 20 | 16
Pain in extremity (Musculoskeletal and connective tissue disorders) | 71 | 61 | 8
Dizziness (Nervous system disorders) | 62 | 50 | 0
Dysgeusia (Nervous system disorders) | 41 | 21 | 0
Headache (Nervous system disorders) | 146 | 77 | 28
Neuropathy peripheral (Nervous system disorders) | 59 | 30 | 16
Paraesthesia (Nervous system disorders) | 31 | 20 | 7
Peripheral sensory neuropathy (Nervous system disorders) | 36 | 27 | 0
Anxiety (Psychiatric disorders) | 31 | 15 | 0
Depression (Psychiatric disorders) | 27 | 30 | 0
Insomnia (Psychiatric disorders) | 69 | 45 | 14
Cough (Respiratory, thoracic and mediastinal disorders) | 100 | 68 | 18
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 61 | 41 | 17
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 121 | 44 | 35
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 24 | 26 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 11
Alopecia (Skin and subcutaneous tissue disorders) | 19 | 25 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 3 | 28 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 17 | 54 | 8
Erythema (Skin and subcutaneous tissue disorders) | 16 | 25 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 18 | 48 | 0
Palmar-Plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 7 | 291 | 7
Pruritus (Skin and subcutaneous tissue disorders) | 32 | 46 | 7
Rash (Skin and subcutaneous tissue disorders) | 64 | 133 | 17
Skin fissures (Skin and subcutaneous tissue disorders) | 2 | 27 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 | 25 | 0
Hypertension (Vascular disorders) | 29 | 11 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.